CLINICAL TRIAL: NCT01757600
Title: Long-term Anatomical and Functional Outcomes of Idiopathic Macular Hole Surgery. The Yield of Spectral-domain OCT Combined With Microperimetry.
Brief Title: Microperimetry and Optical Coherence Tomography (OCT) in Idiopathic Macular Hole
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Principal Investigator, Nicot Frederic, Head of research unit in Ophthalmology department, Centre Hospitalier Universitaire Dijon
Other Study IDs: Arnaud01
Record Dates: First submitted 2012-12-13; First posted 2012-12-31 (Estimated); Last update posted 2012-12-31 (Estimated); Status verified 2012-12

CONDITIONS: Macular Hole
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Macular Hole
  Interventions: Other: Microperimetry

INTERVENTIONS:
Other: Microperimetry

SUMMARY:
To evaluate the correlations between anatomical and functional changes studied with microperimetry (MPM) and spectral-domain OCT (SD-OCT) in patients after successful repair of idiopathic macular hole (MH).

ELIGIBILITY:
Inclusion Criteria:

* Closure of the hole seen on the OCT at 1 year postoperative

Exclusion Criteria:

* Patients with an axial length over 26 mm, diabetes, macular diseases, glaucoma, or postoperative retinal detachment were excluded

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent successful surgery for MH defined as closure of the hole, at least 1 year before.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2010-08; Primary Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Macular sensitivity | 12 months
  To describre mean retinal sensitivity in the 12 and 4 central degrees of the retina in 23 patients one-year after macular hole surgery and thus to correlate macular sensitivities and retinal anatomic features in SD-OCT

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmology Department CHU Dijon, Dijon, Burgundy, France

REFERENCES:
- [Derived] Bonnabel A, Bron AM, Isaico R, Dugas B, Nicot F, Creuzot-Garcher C. Long-term anatomical and functional outcomes of idiopathic macular hole surgery. The yield of spectral-domain OCT combined with microperimetry. Graefes Arch Clin Exp Ophthalmol. 2013 Nov;251(11):2505-11. doi: 10.1007/s00417-013-2339-y. Epub 2013 Apr 26. PMID 23620091